CLINICAL TRIAL: NCT01534442
Title: The Significances of Atropin Administration for the GLP-1 Potentiation of Glucose Induced Insulin Secretion and the Cephalic Insulin Response
Brief Title: Atropin and Glucose Stimulated Insulinsecretion and the Cephalic Insulin Response
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Jonatan I Bagger, MD, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: Atropin clamp
Record Dates: First submitted 2012-02-13; First posted 2012-02-16 (Estimated); Last update posted 2012-12-07 (Estimated); Status verified 2012-12

CONDITIONS: The Focus of This Study is to Evaluete the Significances of the Vagal Cholinerg Nervuos System for the Effect of GLP-1 by Using Atropin Administration.
MeSH Terms: interventions — Atropine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atropin (Active Comparator): Atropin
  Interventions: Drug: Atropine
- Placebo (Placebo Comparator): Saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atropine — 1 mg as a bolus and the and infusion of 80 ng/kg/min for either 105 or 145 minuts.
  Arms: Atropin
Drug: Placebo
  Arms: Placebo

SUMMARY:
The aim of this study is to investigate the role of transmission of vagal cholinerg for the GLP-1 potentiation of the glucose stimulated insulin secretion and the cephalic insulin response by using atropin administration.

The hypothesis is that a great deal of the effects of GLP-1 is mediated via the nervous system and for this reason the investigators will research individuals with an intact nervous supply with and without atropin administration.

DETAILED DESCRIPTION:
GLP-1 is a importent enterogastron and incretin hormone. Rapid degradation of GLP-1 by dipeptidyl peptidase 4 (DPP-4) suggests that GLP-1 may act locally (through vagal afferents) before being degraded. We aimed to clarify the role of vagal innervation on the incretin effect.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 45 years
* normal fasting plasma glucose
* normal hemoglobin
* informed consent

Exclusion Criteria:

* diabetes mellitus
* body mass index above 30
* inflamatoric bowel disease
* intestinal surgery
* serum creatinine above 250 microM
* ALAT above to times normal value
* treatment with medicine wich cannot be paused for 12 hours
* contraindication for treatment with atropin

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
insulin secretion | tree hours
  The insulin secretion during lightly elevated blood glucose during GLP-1 infusions with and without atropin administration is evaluated. Also the insulin secretion during lightly elevated blood glucose during a sham-feeding with and without atropin administration is evaluated.

SECONDARY OUTCOMES:
Plasma PP | 20 time points within tree hours
  20 blood samlpes will be drawn during lightly elevated blood glucose during a sham-feeding with and without atropin administration.
Plasma glucose | 30 within tree hours
  30 blood samlpes will be drawn during lightly elevated blood glucose during a sham-feeding with and without atropin administration.
Plasma GLP-1 | 20 time points within tree hours
  20 blood samlpes will be drawn during lightly elevated blood glucose during a sham-feeding with and without atropin administration.
Plasma GLP-1 | 18 time points within tree hours
  18 blood samples will be drawn during lightly elevated blood glucose during GLP-1 infusions with and without atropin administration.
Plasma GLP-2 | 18 time points within tree hours
  18 blood samples will be drawn during lightly elevated blood glucose during GLP-1 infusions with and without atropin administration.
Plasma GIP | 18 timepoints within tree hours
  18 blood samples will be drawn during lightly elevated blood glucose during GLP-1 infusions with and without atropin administration.
Plasma glucagon | 18 timepoints within tree hours
  18 blood samples will be drawn during lightly elevated blood glucose during GLP-1 infusions with and without atropin administration.
Plasma glucose | 33 timepoints within tree hours
  33 blood samples will be drawn during lightly elevated blood glucose during GLP-1 infusions with and without atropin administration.

CONTACTS AND LOCATIONS:
Overall Officials: Tina Vilsbøll, MD, Dr. med, Study Director — Diabetes research Division, Department of Internal Medicine, Gentofte Hospital, Copenhagen, Denamrk
Locations (2):
- Denmark (2):
  - Diabetes research Division, Department of Internal Medicin, Gentofte Hospital, Hellerup
  - Diabetes Research Division, Department of Internal Medicine, Gentofte Hospital, Copenhagen Denmark, Hellerup

REFERENCES:
- [Derived] Veedfald S, Plamboeck A, Deacon CF, Hartmann B, Knop FK, Vilsboll T, Holst JJ. Cephalic phase secretion of insulin and other enteropancreatic hormones in humans. Am J Physiol Gastrointest Liver Physiol. 2016 Jan 1;310(1):G43-51. doi: 10.1152/ajpgi.00222.2015. Epub 2015 Oct 22. PMID 26492921
- [Derived] Plamboeck A, Veedfald S, Deacon CF, Hartmann B, Vilsboll T, Knop FK, Holst JJ. The role of efferent cholinergic transmission for the insulinotropic and glucagonostatic effects of GLP-1. Am J Physiol Regul Integr Comp Physiol. 2015 Sep;309(5):R544-51. doi: 10.1152/ajpregu.00123.2015. Epub 2015 Jul 1. PMID 26136531